CLINICAL TRIAL: NCT00664274
Title: COMT Genotype and Response to Cognitive Remediation in Schizophrenia
Brief Title: Relation of Catechol-O-methyltransferase (COMT) Genotype and Response to Cognitive Remediation Schizophrenia
Acronym: COMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manhattan Psychiatric Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Clinical Director, Manhattan Psychiatric Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 061/C39-0; 1R03MH078098-01 (NIH); MRPC 2917 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2008-01-10; First posted 2008-04-22 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRT Group (Other)
  Interventions: Behavioral: Cognitive remediation therapy; Genetic: COMT Genotyping

INTERVENTIONS:
Behavioral: Cognitive remediation therapy — 36 sessions of Computerized Cognitive Skills Training, 3 per week for 12 weeks.
  Other Names: educational and behavioral training techniques
Genetic: COMT Genotyping — One time saliva sample is taken to genotype catechol-O-methyltransferase Val158/108Met alleles.
  Other Names: COMT polymorphism; 22q11.21-q11.23

SUMMARY:
This project will explore the relationship between catechol-O-methyltransferase (COMT) Val158/108Met genotype and response to a 12-week computerized neurocognitive rehabilitation (CRT) given to chronic schizophrenic patients.

DETAILED DESCRIPTION:
Cognitive deficits play a crucial role in both the pathogenesis and prognosis of schizophrenia. The COMT gene is functionally expressed in neural systems considered important in a range of healthy brain functions and brain disorders, including schizophrenia. The COMT Met allele has been shown to be associated with a lower activity form of COMT, and with better performance on neurocognitive tests, while the COMT Val allele is associated with poorer executive cognition. This study will investigate the relationship of COMT polymorphism in patients with chronic schizophrenia with the response to CRT targeting visuospatial processing, attention, and cognitive flexibility using MATRICS Consensus Cognitive Battery (MCCB) developed by the NIH-MATRICS initiative.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the active arm of the neurocognitive remediation program
2. Age 18 - 55
3. Inpatients
4. DSM-IV diagnosis of schizophrenia (all subtypes) with illness duration >5 years
5. Auditory and visual acuity adequate to complete cognitive tests
6. Stable dose of oral atypical antipsychotic for at least 4 weeks
7. Total PANSS score > 60
8. RBANS total score ≤ 80
9. MMSE score of greater than or equal to 24
10. Good physical health determined by physical examination, laboratory tests
11. Capacity and willingness to give written informed consent

Exclusion Criteria:

1. Inability to read or speak English
2. Documented disease of the central nervous system
3. History of intellectual impairment pre-dating onset of symptoms of psychosis (e.g. mental retardation)
4. Clinically significant or unstable cardiovascular, renal, hepatic, gastrointestinal, pulmonary or hematologic conditions
5. HIV +
6. Patients diagnosed with substance dependence
7. Currently participating in another experimental study, except for the parent study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2007-04; Primary Completion 2015-01 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of the association of COMT Val108/158 Met genotype with the response to a computerized neurocognitive rehabilitation treatment in patients with chronic schizophrenia. | 12 weeks

SECONDARY OUTCOMES:
To expand the response to a computerized neurocognitive rehabilitation treatment in patients with chronic schizophrenia to other haplotypes or identified genes. | 12 weeks
To assess the differences in demographic variables (e.g. ethnicity, intellectual functioning as measured by WRAT III Reading test, and age) with response to computerized neurocognitive rehabilitation treatment in patients with chronic schizophrenia. | 12 weeks
To assess the differences between antipsychotic treatment and response to computerized neurocognitive rehabilitation treatment in patients with chronic schizophrenia. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, M.D., Principal Investigator — Manhattan Psychiatric Center; Herbert Lachman, M.D., Study Chair — Albert Einstein College of Medicine; Susan Mc Gurk, PhD, Study Chair — New Hampshire-Dartmouth Psychiatric Research Center; Anzalee Khan, PhD, Study Chair — Manhattan Psychiatric Center
Locations (1):
- Manhattan Psychiatric Center, Wards Island, New York, United States

REFERENCES:
- [Background] Woodward ND, Jayathilake K, Meltzer HY. COMT val108/158met genotype, cognitive function, and cognitive improvement with clozapine in schizophrenia. Schizophr Res. 2007 Feb;90(1-3):86-96. doi: 10.1016/j.schres.2006.10.002. Epub 2006 Nov 22. PMID 17123785
- [Background] Bosia M, Bechi M, Marino E, Anselmetti S, Poletti S, Cocchi F, Smeraldi E, Cavallaro R. Influence of catechol-O-methyltransferase Val158Met polymorphism on neuropsychological and functional outcomes of classical rehabilitation and cognitive remediation in schizophrenia. Neurosci Lett. 2007 May 7;417(3):271-4. doi: 10.1016/j.neulet.2007.02.076. Epub 2007 Mar 2. PMID 17383818
- See also: NIMH Press: Brain Scans Reveal How Gene May Boost Schizophrenia Risk — http://www.nimh.nih.gov/science-news/2005/brain-scans-reveal-how-gene-may-boost-schizophrenia-risk.shtml
- See also: Wikipedia: Catechol-O-methyl transferase — http://en.wikipedia.org/wiki/COMT